CLINICAL TRIAL: NCT05328492
Title: Volume Targeted Versus Pressure Targeted Non-invasive Ventilation in Amyotrophic Lateral Sclerosis: a Randomised Control Trial.
Brief Title: Volume Mode Non-invasive Ventilation in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EP545921
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Respiratory Failure; Respiratory Insufficiency; Sleep-Disordered Breathing; Neuro-Degenerative Disease; Neuron Disease, Motor; Nervous System Diseases; Neuromuscular Diseases
Keywords: Non-invasive ventilation; Home ventilation; iVAPS-AE
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Respiratory Insufficiency; Sleep Apnea Syndromes; Motor Neuron Disease; Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iVAPS-AE (Experimental): Patients with ALS and respiratory insufficiency randomised to this arm will be treated with home NIV using the Intelligent Volume-Assured Pressure Support with automatic EPAP (iVAPS-AE) mode.
  Interventions: Device: iVAPS-AE
- ST-mode (Active Comparator): Patients with ALS and respiratory insufficiency randomised to this arm will be treated with home NIV using the spontaneous timed (ST) home NIV mode.
  Interventions: Device: ST-mode

INTERVENTIONS:
Device: iVAPS-AE — Patients randomised to this intervention will commence home NIV in iVAPS-AE mode according to the clinical operating procedures used at the Respiratory and Sleep Science Department. Patients will follow a NHS standard care pathway as described in the study protocol.
  Other Names: ResMed Lumis 150 VPAP ST-A
  Arms: iVAPS-AE
Device: ST-mode — Patients randomised to this intervention will commence home NIV in ST-mode according to the clinical operating procedures used at the Respiratory and Sleep Science Department. Patients will follow a NHS standard care pathway as described in the study protocol.
  Other Names: ResMed Lumis 100 VPAP ST-A
  Arms: ST-mode

SUMMARY:
The purpose of this study is to assess the efficacy of using intelligent volume assured pressure support (iVAPS-AE) versus spontaneous timed (ST) modes of non-invasive ventilation (NIV) in patients diagnosed with amyotrophic lateral sclerosis (ALS).

The investigators believe that the use of iVAPS-AE mode NIV over a 90 day period will produce NIV compliance data and health-related quality of life (HRQOL) scores that are equivalent or no worse compared to ST mode NIV.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is one of five motor neurone diseases (MNDs). It is a rare, incurable disease characterised by progressive destruction of nerve cells called motor neurones that instruct a patient's muscles to contract, to enable all movements, including walking, talking, speaking and swallowing.

Over time as more motor neurone cells are damaged, the muscles used to breathe will weaken and patients will develop breathlessness and sleep disturbances. This can be very distressing and reduce a patient's health- related quality of life (HRQOL). Eventually the condition may progress to the extent that the patient will develop respiratory failure, which is the leading cause of death in ALS.

Respiratory failure is the most frequent cause of death in ALS and as such a significant proportion of ALS cases are complicated by respiratory and bulbar symptoms which can reduce HRQOL from breathlessness, impaired cough and sleep, and can also shorten life expectancy. The use of respiratory support, provided via non-invasive ventilation (NIV), has been shown to be beneficial.

NIV is a safe treatment in ALS and as such current National Institute for Health and Care Excellence (NICE) guidelines recommend a trial of NIV in those ALS patients who develop respiratory impairment

NIV compliance is of significant importance in ALS as it is directly linked to improved survival and health related quality of life. Compliance is affected by various factors including non-invasive ventilation mode, disease type (bulbar vs limb) and baseline physiology.

Various NIV modes exist including pressure support (ST mode) and volume assured pressure support (iVAPS-AE). Evidence suggests that not one mode is more superior, but both have advantages and disadvantages in clinical practice.

This study will follow a standard care pathway and aim to recruit 40 ALS patients randomised to receive ST mode or iVAPS-AE mode. Each patient will enrol onto the study for 90 days and attend 5 hospital visits. The study will assess if iVAPS-AE improves a patient's symptoms sooner and allows a patient to use the NIV for longer periods thereby improving HRQOL.

ELIGIBILITY:
Inclusion Criteria:

Patients with respiratory failure secondary to ALS (diagnosed either at an MND MDT or specialist neurology clinic) according to criteria set out in the NICE guideline (NG42) (2016); Motor neurone disease: assessment and management.

* Patients able to provide informed consent to take part in the research study.
* Patients not contraindicated to commence NIV in accordance with local protocol.
* Patients not currently enrolled in another research study that could alter disease progression.

Exclusion Criteria:

* Acutely unwell or medically complicated patients as assessed by lead investigator. These patients will be urgently reviewed by a dedicated Consultant Physician. The Principal Investigator will be immediately informed.
* An inability to provide informed consent.
* An inability to use NIV.
* Patients whom are contraindicated to commence NIV in accordance with local protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Home NIV Compliance | 90 days
  Measured in hours per night

SECONDARY OUTCOMES:
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) | Baseline, 14, 30, 60, 90 days
  A 12-item questionnaire to monitor the disease progression covering bulbar, motor and respiratory function. Total scores range from 0 to 48. Higher scores indicate better function.
Severe Respiratory Insufficiency Questionnaire (SRI) | Baseline, 14, 30, 60, 90 days
  A 49-item questionnaire to measure health related quality of life in patients receiving long term non-invasive ventilation (NIV). Total scores range from 49 to 245. Higher scores indicate worse outcomes.
Modified Hospital Anxiety and Depression Score (mHADS) | Baseline, 14, 30, 60, 90 days
  A 14-item questionnaire to measure anxiety and depression levels. The questionnaire consists of anxiety sub-scale and depression sub-scale. Scores for each sub-scale range from 0 to 21. Higher scores indicate greater anxiety/depression levels. This version is modified for use in patients diagnosed with amyotrophic lateral sclerosis (ALS).

CONTACTS AND LOCATIONS:
Overall Officials: David G Parr, MD, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Background] Wolf J, Safer A, Wohrle JC, Palm F, Nix WA, Maschke M, Grau AJ. [Causes of death in amyotrophic lateral sclerosis : Results from the Rhineland-Palatinate ALS registry]. Nervenarzt. 2017 Aug;88(8):911-918. doi: 10.1007/s00115-017-0293-3. German. PMID 28184974
- [Background] Goetz CG. Amyotrophic lateral sclerosis: early contributions of Jean-Martin Charcot. Muscle Nerve. 2000 Mar;23(3):336-43. doi: 10.1002/(sici)1097-4598(200003)23:33.0.co;2-l. PMID 10679709
- [Background] Raheja D, Stephens HE, Lehman E, Walsh S, Yang C, Simmons Z. Patient-reported problematic symptoms in an ALS treatment trial. Amyotroph Lateral Scler Frontotemporal Degener. 2016;17(3-4):198-205. doi: 10.3109/21678421.2015.1131831. Epub 2016 Jan 29. PMID 26824413
- [Background] Arnulf I, Similowski T, Salachas F, Garma L, Mehiri S, Attali V, Behin-Bellhesen V, Meininger V, Derenne JP. Sleep disorders and diaphragmatic function in patients with amyotrophic lateral sclerosis. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):849-56. doi: 10.1164/ajrccm.161.3.9805008. PMID 10712332
- [Background] NICE. Recommendations | Motor neurone disease: assessment and management | Guidance | NICE [Internet]. NICE; 2016 [cited 2021 May 10]. Available from: https://www.nice.org.uk/guidance/NG42/chapter/Recommendations#prognostic-factors
- [Background] Ristell HV, Parkes E, Shakespeare J, Bishopp A, Ali A, Parr D. Non-invasive Ventilation Compliance and Survival Trends in Motor Neurone Disease. European Respiratory Journal [Internet]. 2019 Sep 28 [cited 2021 May 5];54(suppl 63). Available from: https://erj.ersjournals.com/content/54/suppl_63/PA3705
- [Background] Nicholson TT, Smith SB, Siddique T, Sufit R, Ajroud-Driss S, Coleman JM 3rd, Wolfe LF. Respiratory Pattern and Tidal Volumes Differ for Pressure Support and Volume-assured Pressure Support in Amyotrophic Lateral Sclerosis. Ann Am Thorac Soc. 2017 Jul;14(7):1139-1146. doi: 10.1513/AnnalsATS.201605-346OC. PMID 28410001
- [Background] Gruis KL, Brown DL, Lisabeth LD, Zebarah VA, Chervin RD, Feldman EL. Longitudinal assessment of noninvasive positive pressure ventilation adjustments in ALS patients. J Neurol Sci. 2006 Aug 15;247(1):59-63. doi: 10.1016/j.jns.2006.03.007. Epub 2006 Apr 24. PMID 16631799
- [Background] Lo Coco D, Marchese S, Pesco MC, La Bella V, Piccoli F, Lo Coco A. Noninvasive positive-pressure ventilation in ALS: predictors of tolerance and survival. Neurology. 2006 Sep 12;67(5):761-5. doi: 10.1212/01.wnl.0000227785.73714.64. Epub 2006 Aug 9. PMID 16899545
- [Background] Kim SM, Park KS, Nam H, Ahn SW, Kim S, Sung JJ, Lee KW. Capnography for assessing nocturnal hypoventilation and predicting compliance with subsequent noninvasive ventilation in patients with ALS. PLoS One. 2011 Mar 30;6(3):e17893. doi: 10.1371/journal.pone.0017893. PMID 21479202
- [Background] Mansell SK, Cutts S, Hackney I, Wood MJ, Hawksworth K, Creer DD, Kilbride C, Mandal S. Using domiciliary non-invasive ventilator data downloads to inform clinical decision-making to optimise ventilation delivery and patient compliance. BMJ Open Respir Res. 2018 Mar 3;5(1):e000238. doi: 10.1136/bmjresp-2017-000238. eCollection 2018. PMID 29531743
- [Background] Rudnicki SA, Andrews JA, Bian A, Cockroft BM, Cudkowicz ME, Hardiman O, Malik FI, Meng L, Wolff AA, Shefner JM; VITALITY-ALS STUDY GROUP. Noninvasive ventilation use by patients enrolled in VITALITY-ALS. Amyotroph Lateral Scler Frontotemporal Degener. 2021 Nov;22(7-8):486-494. doi: 10.1080/21678421.2021.1904993. Epub 2021 Apr 1. PMID 33792451
- [Background] Vitacca M, Banfi P, Montini A, Paneroni M. Does timing of initiation influence acceptance and adherence to NIV in patients with ALS? Pulmonology. 2020 Jan-Feb;26(1):45-48. doi: 10.1016/j.pulmoe.2019.05.007. Epub 2019 Jun 5. PMID 31175073
- [Background] Kleopa KA, Sherman M, Neal B, Romano GJ, Heiman-Patterson T. Bipap improves survival and rate of pulmonary function decline in patients with ALS. J Neurol Sci. 1999 Mar 15;164(1):82-8. doi: 10.1016/s0022-510x(99)00045-3. PMID 10385053
- [Background] Czudaj KP, Suchi S, Schonhofer B. [Physiological parameters of breathing and the impact of non-invasive ventilation (NIV) on patients with amyotrophic lateral sclerosis (ALS)]. Pneumologie. 2009 Dec;63(12):687-92. doi: 10.1055/s-0029-1215130. Epub 2009 Nov 3. German. PMID 19890778
- [Background] Bach JR. Amyotrophic lateral sclerosis. Communication status and survival with ventilatory support. Am J Phys Med Rehabil. 1993 Dec;72(6):343-9. PMID 8260126
- [Background] Pinto AC, Evangelista T, Carvalho M, Alves MA, Sales Luis ML. Respiratory assistance with a non-invasive ventilator (Bipap) in MND/ALS patients: survival rates in a controlled trial. J Neurol Sci. 1995 May;129 Suppl:19-26. doi: 10.1016/0022-510x(95)00052-4. PMID 7595610
- [Background] Rabec C, Rodenstein D, Leger P, Rouault S, Perrin C, Gonzalez-Bermejo J; SomnoNIV group. Ventilator modes and settings during non-invasive ventilation: effects on respiratory events and implications for their identification. Thorax. 2011 Feb;66(2):170-8. doi: 10.1136/thx.2010.142661. Epub 2010 Oct 14. PMID 20947891
- [Background] Sancho J, Servera E, Morelot-Panzini C, Salachas F, Similowski T, Gonzalez-Bermejo J. Non-invasive ventilation effectiveness and the effect of ventilatory mode on survival in ALS patients. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Mar;15(1-2):55-61. doi: 10.3109/21678421.2013.855790. Epub 2013 Nov 25. PMID 24266679
- [Background] Morelot-Panzini C, Bruneteau G, Gonzalez-Bermejo J. NIV in amyotrophic lateral sclerosis: The 'when' and 'how' of the matter. Respirology. 2019 Jun;24(6):521-530. doi: 10.1111/resp.13525. Epub 2019 Mar 25. PMID 30912216